CLINICAL TRIAL: NCT02630641
Title: Impact of the Perception of Cohesion Within a Relationship (Dyadic Adjustment) on the Quality of Life of Patients With Prostate Cancer With Gonadotropin-releasing Hormone (GnRH) Agonist Therapy Initiated by the Urologist in the Routine Practice. Evaluation by the Patient and the Partner.
Brief Title: Perception of Cohesion Within a Relationship (Dyadic Adjustment) on the Quality of Life of Patients With Prostate Cancer With Gonadotropin-releasing Hormone.
Acronym: EQUINOXE
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-54-52014-218
Record Dates: First submitted 2015-12-11; First posted 2015-12-15 (Estimated); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prostate cancer patients
  Interventions: Drug: Gonadotropin-releasing Hormone (GnRH) agonist therapy

INTERVENTIONS:
Drug: Gonadotropin-releasing Hormone (GnRH) agonist therapy — This is a non-interventional study. Thus, investigators are free to choose GnRH agonist therapy product, and modalities of administration in accordance with local Summary of Product Characteristics.

SUMMARY:
The general hypothesis put forward in this study is that the degree of cohesion (agreement) in the relationship, or dyadic adjustment affects a patient's quality of life and clinical course during the first few critical months following diagnosis and the introduction of treatment. The level of cohesion in the relationship is certainly not the only parameter associated with changes in the quality of life. Other factors must also be investigated such as level of education, circumstances surrounding the diagnosis (new diagnosis or relapse), management (single therapy or adjuvant therapy), the level of physical activity, the patient's age and the presence of functional disorders, etc.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting with histologically confirmed prostate cancer.
* Patient eligible to start GnRH agonist therapy, either as monotherapy or adjuvant therapy, and for whom one of these treatments was selected voluntarily by the urologist, prior to the start of the study.
* Patient currently living with the same partner for at least 6 months.
* Patient and partner capable of reading, understanding and returning an evaluation self-questionnaire 6 months after the initial consultation.
* Patient giving its written consent to participate to the study.

Exclusion Criteria:

* The subject is participating in another clinical trial.
* Patient who has received a GnRH agonist therapy during the last 2 years.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prostate cancer patients and their partners recruited by urologists.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2015-10; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change in quality of life of the patient. | Baseline and 6 months
  Assessment of the dyadic adjustment and its impact on the quality of life of the patient through self-questionnaire by the patient and the partner

SECONDARY OUTCOMES:
Assessment of representations of illness | Baseline
  Self-questionnaire by the patient and the partner
Correlations between quality of life specific to prostate cancer, general quality of life and dyadic adjustment. | 6 months
  Self-questionnaire by the patient only
Proportion of couples with a consistency or inconsistency level of dyadic adjustment | 6 months
Investigation of factors associated with patient's perception of dyadic adjustment on changes quality of life | Baseline and 6 months
  Self-questionnaire by the patient and the partner

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Ipsen Central Contact, Paris, France

REFERENCES:
- [Result] Droupy S, Colson MH, Pello-Leprince-Ringuet N, Perrot V, Descazeaud A. EQUINOXE study: Impact of relational cohesion and sexuality on the quality of life of patients treated with gonadotropin-releasing hormone agonist for prostate cancer. BJUI Compass. 2021 Oct 19;3(1):45-54. doi: 10.1002/bco2.92. eCollection 2022 Jan. PMID 35475155